CLINICAL TRIAL: NCT02667613
Title: Effet de la réadaptation Sur Les déficiences, Limitations d'activité et Restriction de la Participation Des Enfants présentant Des lésions Neurologiques Non-évolutives. Part IIb
Brief Title: Changes in Everydaylife Activity of Children With CP During HABIT-ILE
Acronym: change_CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B403201316810b
Record Dates: First submitted 2015-12-21; First posted 2016-01-29 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
Keywords: motor skill learning; functional changes; neuroplastic changes
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HABIT-ILE (Experimental): HABIT-ILE (Hand and arm bimanual intensive therapy including lower extremities) will be applied over 2 weeks.
  Interventions: Other: HABIT-ILE
- Control (Active Comparator): A two weeks period of usual customary care.
  Interventions: Other: Control

INTERVENTIONS:
Other: HABIT-ILE — Hand and arm bimanual intensive therapy including lower extremities
  Arms: HABIT-ILE
Other: Control — Usual customary care
  Arms: Control

SUMMARY:
Studying in a RCT the changes in everyday llife activities of children with CP during HABIT-ILE or control period, changes being scored by parents and by experts.

DETAILED DESCRIPTION:
Studying in a RCT the changes in everyday llife activities of children with CP (unilateral and bilateral) during HABIT-ILE or control period, changes being scored by parents and by experts on ABILHAND-Kids, the PEDI, the ACTIVLM-CP and the COPM. Investigate neuroplastic changes and correlation with everyday life changes.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* ability to make a few steps with a walking device
* ability to pick a light object from a table with the more affected hand
* ability to understand simple games

Exclusion Criteria:

* no active seizure
* no botulinum toxin in the 6 months previous to the intervention or during intervention time
* major visual deficit

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in activity measure (questionnaires) | 2 weeks of intervention and 4 months (follow-up)
  change in a measure of daily activities through ABILHAND-Kids, ACTIVLIM-CP and the COPM

SECONDARY OUTCOMES:
neuroplastic changes in the cortex (MRI, fMRI, DTI, TMS) | baseline and 2 weeks of intervention
  measure of neuroplastic changes through TMS and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, PhD, Principal Investigator — Institute of Neuroscience, Université catholique de Louvain
Locations (1):
- Institute of Neuroscience, Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Araneda R, Dricot L, Ebner-Karestinos D, Paradis J, Gordon AM, Friel KM, Bleyenheuft Y. Brain activation changes following motor training in children with unilateral cerebral palsy: An fMRI study. Ann Phys Rehabil Med. 2021 May;64(3):101502. doi: 10.1016/j.rehab.2021.101502. Epub 2021 Mar 22. PMID 33647530
- [Derived] Bleyenheuft Y, Dricot L, Ebner-Karestinos D, Paradis J, Saussez G, Renders A, De Volder A, Araneda R, Gordon AM, Friel KM. Motor Skill Training May Restore Impaired Corticospinal Tract Fibers in Children With Cerebral Palsy. Neurorehabil Neural Repair. 2020 Jun;34(6):533-546. doi: 10.1177/1545968320918841. Epub 2020 May 14. PMID 32407247
- [Derived] Paradis J, Dispa D, De Montpellier A, Ebner-Karestinos D, Araneda R, Saussez G, Renders A, Arnould C, Bleyenheuft Y. Interrater Reliability of Activity Questionnaires After an Intensive Motor-Skill Learning Intervention for Children With Cerebral Palsy. Arch Phys Med Rehabil. 2019 Sep;100(9):1655-1662. doi: 10.1016/j.apmr.2018.12.039. Epub 2019 Feb 18. PMID 30790557